CLINICAL TRIAL: NCT06921512
Title: TCM Daoyin for Anxiety and Depression Symptoms: Psychological Effects and Biological Mechanisms
Brief Title: TCM Daoyin for Anxiety/Depression: Psychological Effects and Biological Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Lu Ying, MM, assistant researcher, Shanghai University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24KFL060
Record Dates: First submitted 2025-03-31; First posted 2025-04-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Symptom; Depression Symptom
Keywords: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is a single-arm trial with 20 participants undergoing a 12-week TCM Daoyin exercise intervention (2 sessions per week), followed by a 12-week observational follow-up period. Primary outcomes (HAMA-14 and HAMD-17 scores) and exploratory biomarkers (inflammatory markers, immune cell subsets, and serum metabolomics) will be assessed at baseline, 12 weeks, and 24 weeks. No control group is included.
Masking Description: This is an open-label, single-arm trial. While no formal masking is applied, the outcomes assessor will not have access to participant adherence records or follow-up exercise engagement data to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCM Daoyin Exercise Group (Experimental): Participants will receive a 12-week TCM Daoyin training program led by qualified physicians. Structured group sessions will incorporate movement regulation, breath regulation, and mind regulation to alleviate anxiety and depression symptoms.
  Interventions: Behavioral: TCM Daoyin exercise

INTERVENTIONS:
Behavioral: TCM Daoyin exercise — Participants will receive a 12-week, group-based TCM Daoyin intervention consisting of two 90-minute sessions per week (total: 24 sessions), led by qualified physicians. Each session integrates movement regulation, breath regulation, and mind regulation, aiming to alleviate anxiety and depression symptoms. Each session includes a 10-minute warm-up and a 10-minute cool-down.
  Compliance and Analysis:
  Per-protocol analysis will include participants who attend ≥80% of sessions (≥19/24 sessions). Safety analyses will be conducted on all enrolled participants (n=20) following the intention-to-treat (ITT) principle.

SUMMARY:
This 12-week single-arm clinical trial investigates the effects of Traditional Chinese Medicine (TCM) Daoyin exercise on anxiety and depression symptoms in 20 participants, followed by a 12-week observational follow-up period.

The primary outcome is the change in Hamilton Anxiety Rating Scale (HAMA-14) and Hamilton Depression Rating Scale (HAMD-17) scores at 12 weeks. A secondary outcome will assess these scores at 24 weeks to evaluate sustained effects. Additional secondary outcomes include the Depression, Anxiety, and Stress Scale (DASS-21) and Pittsburgh Sleep Quality Index (PSQI) to further assess changes in mood and sleep quality at the same time points.

Exploratory analyses will examine inflammatory markers, immune cell subsets, serum metabolomics, and gut microbiota at baseline, 12 weeks, and 24 weeks to identify potential biological correlates. During the follow-up period, participants will record their actual exercise engagement, allowing investigators to explore long-term associations. Findings may provide insights for future mechanistic studies on TCM's role in mental health.

DETAILED DESCRIPTION:
Anxiety and depression are among the most prevalent mental health conditions and are commonly associated with inflammation, immune dysregulation, and metabolic disturbances. Traditional Chinese Medicine (TCM) interventions, such as Daoyin exercise-a form of guided movement and breathing-have historically been used to promote mental well-being. However, their biological mechanisms remain inadequately understood.

This 12-week, single-arm clinical trial aims to evaluate the effects of a structured Daoyin exercise program on subclinical anxiety and depression symptoms in 20 adult participants. After completing the 12-week intervention, participants will enter a 12-week observational follow-up period, during which they may choose to continue or discontinue the practice at their discretion. Actual exercise engagement during the follow-up will be self-recorded using daily logs.

The primary outcome is the change in Hamilton Anxiety Rating Scale (HAMA-14) and Hamilton Depression Rating Scale (HAMD-17) scores from baseline to 12 weeks. A secondary outcome will assess the persistence of these effects at 24 weeks. Additional psychological assessments include the Depression, Anxiety, and Stress Scale (DASS-21) and the Pittsburgh Sleep Quality Index (PSQI), evaluated at baseline, 12 weeks, and 24 weeks to assess broader changes in mood and sleep quality.

Exploratory outcomes will investigate potential biological mechanisms by measuring:

* Inflammatory markers (e.g., interleukin-10 [IL-10], interleukin-6 [IL-6], tumor necrosis factor-alpha [TNF-α]) via serum ELISA
* Immune cell subsets (e.g., cluster of differentiation 3-positive [CD3+], cluster of differentiation 4-positive [CD4+], cluster of differentiation 8-positive [CD8+] T cells) via flow cytometry
* Serum metabolomics using liquid chromatography-mass spectrometry (LC-MS) to identify metabolic changes potentially related to the effects of Daoyin exercise on anxiety and depression
* Gut microbiota composition using high-throughput sequencing techniques

Samples will be collected at baseline, 12 weeks, and 24 weeks. These data will help identify physiological pathways potentially linked to improvements in anxiety and depression symptoms.

Participants will be included based on clinician assessment and confirmed subclinical symptoms, with HAMA-14 scores between 14-29 and HAMD-17 scores between 7-14, without meeting ICD-10 diagnostic criteria for anxiety or depressive disorders. All psychological and biological evaluations will occur at three time points: baseline, post-intervention (12 weeks), and follow-up (24 weeks).

The results may offer preliminary evidence for integrating Daoyin exercise into mental health self-management strategies and provide a foundation for future research into TCM's biological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Primary symptoms of anxiety and depression, with a Hamilton Anxiety Rating Scale (HAMA-14) score between 14 and 29 and a Hamilton Depression Rating Scale (HAMD-17) score between 7 and 14.
* No prior use of psychotropic medication, or at least six months since discontinuation.
* Aged 18 to 65 years (male or female).
* Clear consciousness and normal cognitive function, with the ability to communicate effectively, read, express thoughts, and engage in daily activities independently.
* Willing and able to comply with blood and stool sample collection.
* Voluntary participation, with signed informed consent provided before enrollment.

Exclusion Criteria:

* Diagnosed anxiety disorder or depressive disorder based on ICD-10 criteria.
* Bipolar disorder, psychotic disorders (e.g., schizophrenia), or organic mental disorders (e.g., Alzheimer's disease).
* History of alcohol or substance use disorder within the past year, current psychiatric medication use, or high suicide risk.
* Severe or unstable medical conditions, including immune or endocrine disorders or other serious illnesses.
* Physical or psychological limitations preventing participation in the TCM Daoyin intervention.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
14-item Hamilton Anxiety Rating Scale (HAMA-14) | Change from Baseline at 12 weeks
  The 14-item Hamilton Anxiety Rating Scale (HAMA-14) is a clinician-rated assessment (structured interview) of patients' anxiety symptoms. The scale evaluates symptoms experienced over the past 7 days, with higher cumulative scores indicating more severe anxiety.
  Each item is rated on a 5-point scale from 0 (no symptoms) to 4 (very severe symptoms). The total score ranges from 0 to 56, with severity levels categorized as follows:
  * ≥29: Severe anxiety disorder
  * 21-28: Marked anxiety disorder
  * 14-20: Anxiety disorder
  * 8-13: Suspected anxiety disorder
  * ≤7: No anxiety disorder
17-item Hamilton Depression Rating Scale (HAMD-17) | Change from Baseline at 12 weeks
  The 17-item Hamilton Depression Rating Scale (HAMD-17) is a clinician-rated assessment (structured interview) of patients' depressive symptoms. The scale assesses symptoms over the past 7 days, with higher cumulative scores indicating more severe depression.
  Each item is rated on a 5-point scale from 0 (no symptoms) to 4 (very severe symptoms). The total score ranges from 0 to 52, with severity levels categorized as follows:
  * ≥25: Severe depression disorder
  * 18-24: Moderate depression
  * 13-17: Mild depression disorder
  * 8-12: Suspected depression disorder
  * ≤7: No depression disorder

SECONDARY OUTCOMES:
14-item Hamilton Anxiety Rating Scale (HAMA-14) | Change from 12 weeks to 24 weeks
  The 14-item Hamilton Anxiety Rating Scale (HAMA-14) is a clinician-rated assessment (structured interview) of patients' anxiety symptoms. The scale evaluates symptoms experienced over the past 7 days, with higher cumulative scores indicating more severe anxiety.
  Each item is rated on a 5-point scale from 0 (no symptoms) to 4 (very severe symptoms). The total score ranges from 0 to 56, with severity levels categorized as follows:
  * ≥29: Severe anxiety disorder
  * 21-28: Marked anxiety disorder
  * 14-20: Anxiety disorder
  * 8-13: Suspected anxiety disorder
  * ≤7: No anxiety disorder
14-item Hamilton Anxiety Rating Scale (HAMA-14) | Change from Baseline to 24 weeks
  The 14-item Hamilton Anxiety Rating Scale (HAMA-14) is a clinician-rated assessment (structured interview) of patients' anxiety symptoms. The scale evaluates symptoms experienced over the past 7 days, with higher cumulative scores indicating more severe anxiety.
  Each item is rated on a 5-point scale from 0 (no symptoms) to 4 (very severe symptoms). The total score ranges from 0 to 56, with severity levels categorized as follows:
  * ≥29: Severe anxiety disorder
  * 21-28: Marked anxiety disorder
  * 14-20: Anxiety disorder
  * 8-13: Suspected anxiety disorder
  * ≤7: No anxiety disorder
17-item Hamilton Depression Rating Scale (HAMD-17) | Change from 12 weeks to 24 weeks
  The 17-item Hamilton Depression Rating Scale (HAMD-17) is a clinician-rated assessment (structured interview) of patients' depressive symptoms. The scale assesses symptoms over the past 7 days, with higher cumulative scores indicating more severe depression.
  Each item is rated on a 5-point scale from 0 (no symptoms) to 4 (very severe symptoms). The total score ranges from 0 to 52, with severity levels categorized as follows:
  * ≥25: Severe depression disorder
  * 18-24: Moderate depression
  * 13-17: Mild depression disorder
  * 8-12: Suspected depression disorder
  * ≤7: No depression disorder
17-item Hamilton Depression Rating Scale (HAMD-17) | Change from Baseline to 24 weeks
  The 17-item Hamilton Depression Rating Scale (HAMD-17) is a clinician-rated assessment (structured interview) of patients' depressive symptoms. The scale assesses symptoms over the past 7 days, with higher cumulative scores indicating more severe depression.
  Each item is rated on a 5-point scale from 0 (no symptoms) to 4 (very severe symptoms). The total score ranges from 0 to 52, with severity levels categorized as follows:
  * ≥25: Severe depression disorder
  * 18-24: Moderate depression
  * 13-17: Mild depression disorder
  * 8-12: Suspected depression disorder
  * ≤7: No depression disorder
The Depression, Anxiety, and Stress Scale-21 (DASS-21) | Change from Baseline at 6 weeks, 12 weeks, 18 weeks, and 24 weeks.
  The DASS-21 is a self-reported assessment used to measure the severity of depression, anxiety, and stress symptoms experienced by individuals over the past week. Higher cumulative scores on each subscale indicate more severe symptoms of depression, anxiety, or stress. The DASS-21 includes three subscales, each with 7 items: one for depression, one for anxiety, and one for stress. Each item is rated on a 4-point scale ranging from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time).
  Subscale scores are calculated by summing the responses to the seven items in each subscale and multiplying the total by 2. The following cutoff values are used to categorize symptom severity:
  * Depression: A score greater than 9 indicates mild to severe depression.
  * Anxiety: A score greater than 7 indicates mild to severe anxiety.
  * Stress: A score greater than 14 indicates mild to severe stress.
Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline at 6 weeks, 12 weeks, 18 weeks, and 24 weeks.
  The PSQI consists of 19 self-rated items and 5 items rated by a roommate or bed partner. The 19th self-rated item and the 5 items rated by others are not included in the scoring. The remaining 18 self-rated items are grouped into 7 components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored from 0 to 3, with higher scores indicating worse sleep quality. The total score is the sum of the 7 components, with a range of 0 to 21. It is used to assess the participant's subjective sleep quality over the past month, where higher scores indicate poorer sleep quality.
Changes in Inflammatory Markers | Change from Baseline at 12 weeks and 24 weeks
  Changes in inflammatory markers (e.g., interleukin-10 [IL-10], interleukin-6 [IL-6], tumor necrosis factor-alpha [TNF-α]) from baseline to 12 weeks and 24 weeks to explore the potential biological mechanisms underlying the effects of Daoyin exercise on anxiety and depression.
Changes in Immune Cell Subsets | Change from Baseline at 12 weeks and 24 weeks
  Changes in immune cell subsets (e.g., cluster of differentiation 3-positive [CD3+], cluster of differentiation 4-positive [CD4+], cluster of differentiation 8-positive [CD8+] T cells) from baseline to 12 weeks and 24 weeks to explore the potential biological mechanisms underlying the effects of Daoyin exercise on anxiety and depression.
Changes in Serum Metabolomics | Change from Baseline at 12 weeks and 24 weeks
  Changes in serum metabolomics from baseline to 12 weeks and 24 weeks to explore the potential biological mechanisms underlying the effects of Daoyin exercise on anxiety and depression.
Changes in Gut Microbiota | Change from Baseline at 12 weeks and 24 weeks
  Changes in gut microbiota from baseline to 12 weeks and 24 weeks to explore the potential biological mechanisms underlying the effects of Daoyin exercise on anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, Master, Principal Investigator — Shanghai Qigong Research Institute
Locations (1):
- Shanghai Qigong Research Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: No